CLINICAL TRIAL: NCT01681459
Title: Effects of Lipids on Gastric Emptying, Satiety Hormones, and Appetite in Severe Overweight
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Jan Lysgaard Madsen, Chief Physician, MD, DMSci, Hvidovre University Hospital
Other Study IDs: H-4-2011-060
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Effects of Lipids on Gastric Emptying; Effects of Lipids on Satiety Hormones; Effects of Lipids on Appetite
Keywords: Free fatty acid; Triglyceride; Gastric emptying; Satiety hormones; Appetite; Severe obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In lean subjects, free fatty acid (FFA) promotes gut hormone release, delays gastric emptying, and reduces appetite and energy intake more than an isocaloric load of triglyceride (TG). In obesity, the gastrointestinal sensitivity to food components may be reduced. In this study, the investigators compare the effects of the FFA oleic acid and the TG olive oil on gut hormone secretion, gastric emptying, appetite sensation, and subsequent energy intake in lean and severely obese subjects.

DETAILED DESCRIPTION:
Nutritional lipid within the lumen of small intestine causes a range of physiological responses that suppress appetite and reduce energy intake. Thus, intestinal fat promotes the release of gastrointestinal hormones such as cholecystokinin (CCK), peptide-YY (PYY) and glucagon-like peptide-1 (GLP-1) that modulate gastrointestinal motility and are important for appetite regulation and food consumption.

The effect of ingested fat on gut hormone secretion is highly dependent on the lipolysis of triglycerides (TGs) into free fatty acids (FFAs). It has been demonstrated that adding a lipase inhibitor (tetrahydrolipstatin) to a pure fat meal accelerates gastric emptying and reduces CCK release. Furthermore, administration of tetrahydrolipstatin with an intraduodenal infusion of TG attenuates gastric relaxation and antro-pyloro-duodenal motility and reduces the release of CCK, PYY, and GLP-1 compared to TG alone. Finally, intragastric administration of FFA delays gastric emptying and augments the release of CCK and PYY compared to an isocaloric administration of TG. Hence, the presence of FFAs more than TGs within the small intestine seem to play a pivotal role in the regulation of appetite and energy intake.

Whereas acute intake of FFA represents a potent stimulus for suppression of appetite and energy intake, epidemiological evidence relates long-term high dietary fat intake with obesity and it is known that obese individuals prefer food with high fat content. The mechanisms behind this paradox remain unclear. However, sustained high fat-diet may change gastromotor responses and gut hormonal release to a dietary load of lipids. Moreover intraduodenal sensitivity to FFA (oleic acid) was recently reported to be reduced in obese subjects. The reduced appetite and energy intake after FFAs compared to TGs may, therefore, not apply to obese subjects.

The aims of this study are to evaluate gastric emptying, gut hormone secretion, appetite sensation, and energy intake after isocaloric gastric administration of FFA (oleic acid) and TG (olive oil) in lean and severely obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Lean subjects: BMI 20-25
* Severely obese subjects: BMI > 50

Exclusion Criteria:

-Gastrointestinal symptoms

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 lean subjects and 10 severely obese subjects
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark